CLINICAL TRIAL: NCT00401492
Title: Phase II Study of Chemotherapy With Gemcitabine in Prolonged Infusion or With Schedules With Cisplatin in Non-small Cell Lung Cancer Elderly Patients
Brief Title: MILES-02: Study of Chemotherapy Treatment and Toxicity in Elderly Patients With Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MILES-02
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: elderly; chemotherapy; quality of life; ADL; toxicity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Vinorelbine

INTERVENTIONS:
Drug: gemcitabine prolonged continuous infusion
Drug: cisplatin
Drug: vinorelbine

SUMMARY:
The main purpose of this study is to describe activity and toxicity of single-agent gemcitabine given as prolonged infusion, and of two 2-drug combinations containing cisplatin (cisplatin + vinorelbine, and cisplatin + gemcitabine) in the treatment of elderly patients with advanced non small cell lung cancer

DETAILED DESCRIPTION:
The study design includes three parallel phase II studies, all with the same rules for patient selection and outcome assessment. In the two studies of cisplatin-based doublets, a dose-finding phase is planned, with subsequent cohorts of 6 patients treated with increasing doses of cisplatin (50-60-70 mg/m²). Following this phase, patients will be assigned to the three studies through a randomization procedure, to reduce selection biases.

Arm A: gemcitabine:

Gemcitabine 1200 mg/m2 intravenously in 2 hours (10 mg/m²/minute) on days 1 & 8 of each cycle, every 21 days, for a maximum of 6 cycles.

Arm B: cisplatin + vinorelbine:

Vinorelbine 25 mg/m² on days 1 & 8, followed by Cisplatin (50 or 60 or 70 mg/m²) on day 1 of each cycle, every 21 days, for a maximum of 6 cycles.

Arm C: cisplatin + gemcitabine:

Gemcitabine 1000 mg/m2,, on days 1 & 8, followed by Cisplatin (50 or 60 or 70 mg/m²) on day 1 of each cycle, every 21 days, for a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of NSCLC
* Stage IV or IIIB with pleural effusion or metastatic supraclavicular lymphoadenopathy
* Age > o = 70 years.
* Written informed consent.

Exclusion Criteria:

* Performance status (ECOG) ³2
* Previous chemotherapy.
* Symptomatic brain metastases requiring synchronous radiotherapy
* Previous radiotherapy (completed less than 4 weeks before enrollment)
* Previous or synchronous malignant disease (except adequately treated non melanomatous skin cancer or carcinoma in situ of the cervix) if diagnosed in the last five years before enrollment.
* Neutrophils < 2.000/mm³ or platelets < 100.000/mm³ or hemoglobin < 10 g/dl.
* Serum creatinine > 1.5 times the UNL.
* GOT and/or GPT >1.25 times the UNL or serum total bilirubin >1.25 times the UNL without hepatic metastases.
* GOT and/or GPT >2.5 times the UNL or serum total bilirubin >1.5 times the UNL with hepatic metastases.
* Other concomitant diseases contraindicating the study treatments.
* Refusal of written informed consent.
* Follow-up impossible.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 159 (Actual)
Dates: Start 2002-06; Primary Completion 2006-12 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Activity and toxicity of monochemotherapy with gemcitabine as prolonged infusion
Toxicity and activity of 2 standard polychemotherapy cisplatin based treatments (cisplatin and vinorelbine , and cisplatin and gemcitabine

SECONDARY OUTCOMES:
patient quality of life
the prognostic significance of the ADL and IADL scales for time to progression and survival
exploratory predictive clinical variables for chemotherapy related toxicity
exploratory predictive clinical variables for response to chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — San Giuseppe Moscati Hospital; Francesco Perrone, M.D., Principal Investigator — National Cancer Institute, Naples Italy

REFERENCES:
- [Result] Gridelli C, Maione P, Illiano A, Piantedosi FV, Favaretto A, Bearz A, Robbiati SF, Filipazzi V, Lorusso V, Carrozza F, Iaffaioli RV, Manzione L, Gallo C, Morabito A, Perrone F. Cisplatin plus gemcitabine or vinorelbine for elderly patients with advanced non small-cell lung cancer: the MILES-2P studies. J Clin Oncol. 2007 Oct 10;25(29):4663-9. doi: 10.1200/JCO.2007.12.5708. PMID 17925563
- [Result] Gridelli C, De Maio E, Barbera S, Sannicolo M, Piazza E, Piantedosi F, Brancaccio L, Morabito A, Maione P, Renda F, Signoriello G, Perrone F; MILES Investigators. The MILES-2G phase 2 study of single-agent gemcitabine with prolonged constant infusion in advanced non-small cell lung cancer elderly patients. Lung Cancer. 2008 Jul;61(1):67-72. doi: 10.1016/j.lungcan.2007.12.002. PMID 18683299